CLINICAL TRIAL: NCT01700686
Title: The Effect of Gastric Bypass Surgery on Gut Hormones Related to Bone Remodeling and Intestinal Growth.
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Bolette Hartmann, PhD, University of Copenhagen
Other Study IDs: GBPK
Record Dates: First submitted 2012-10-02; First posted 2012-10-04 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Bone Loss
MeSH Terms: conditions — Obesity; Bone Diseases, Metabolic | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples are retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese subjects: Meal test and dexa scan
  Interventions: Other: Meal test and dexa scan

INTERVENTIONS:
Other: Meal test and dexa scan — Body composition is determined by whole body deca scan and bone mineral density is determined dy dexa scans of the lumbar spine and the proximal femur.

SUMMARY:
The overall purpose is to explore the link between the gut and the bones by investigating meal stimulated changes in the blood level of a number of hormones and markers related to intestinal growth and bone turnover in patients undergoing surgery for obesity (gastric bypass). The hormones will be measured in blood samples taken before and after surgery. The results are compared with changes in body weight and body composition as measured by DEXA scanning.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians fulfilling the criteria for laparoscopic gastric bypass.
* BMI>40kg/m2.

Exclusion Criteria:

* Pregnancy
* Chronic obstructive pulmonary disease
* Diabetes mellitus
* Chronic inflammatory bowel disease
* Major psychiatric disorder
* Drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are recruited from The Bariatric Clinic, The Hospital of Roskilde-Koege, The University of Copenhagen.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Meal stimulated changes in gut hormones and bone markers. | Before surgery and 4 weeks and 6 months after surgery.

SECONDARY OUTCOMES:
Changes in bone mass and body composition. | Before surgery and 6 months after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Bolette Hartmann, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- Hospital of Roskilde-Koege, The University of Copenhagen, Koege, Denmark